CLINICAL TRIAL: NCT04516447
Title: A Phase 1b Study of ZN-c3 in Combination With Chemotherapy or Bevacizumab in Subjects With Ovarian, Peritoneal, or Fallopian Tube Cancer
Brief Title: A Study of ZN-c3 in Patients With Ovarian Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: K-Group, Beta, Inc., a wholly owned subsidiary of Zentalis Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZN-c3-002
Record Dates: First submitted 2020-08-11; First posted 2020-08-18 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Solid Tumor; Epithelial Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: Solid Tumor
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — Drug Evaluation; Carboplatin; liposomal doxorubicin; Paclitaxel; Gemcitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Combination with carboplatin (Experimental): combined with azenosertib
  Interventions: Drug: ZN-c3; Drug: Carboplatin
- Combination with PLD (Experimental): combined with azenosertib
  Interventions: Drug: ZN-c3; Drug: Pegylated liposomal doxorubicin
- Combination with paclitaxel (Experimental): combined with azenosertib
  Interventions: Drug: ZN-c3; Drug: Paclitaxel
- Combination with gemcitabine (Experimental): combined with azenosertib
  Interventions: Drug: ZN-c3; Drug: Gemcitabine
- Combination with bevacizumab (Experimental): combined with azenosertib
  Interventions: Drug: ZN-c3; Biological: Bevacizumab

INTERVENTIONS:
Drug: ZN-c3 — Investigational drug
  Other Names: Study drug; Azenosertib
Drug: Carboplatin — Carboplatin is an approved drug
  Arms: Combination with carboplatin
Drug: Pegylated liposomal doxorubicin — Pegylated liposomal doxorubicin (PLD) is an approved drug
  Arms: Combination with PLD
Drug: Paclitaxel — Paclitaxel is an approved drug
  Arms: Combination with paclitaxel
Drug: Gemcitabine — Gemcitabine is an approved drug
  Arms: Combination with gemcitabine
Biological: Bevacizumab — Combined with azenosertib
  Arms: Combination with bevacizumab

SUMMARY:
This is a Phase 1b open-label, multicenter study, evaluating the safety, tolerability, preliminary clinical activity, pharmacokinetics (PK), and pharmacodynamics of ZN-c3 in combination with other drugs.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed high-grade serous epithelial ovarian carcinoma, fallopian tube, or peritoneal carcinoma.
* Subjects must have received 1 or 2 prior therapeutic regimens/lines of therapy in the advanced or metastatic setting.
* Measurable disease per RECIST version 1.1.
* Adequate hematologic and organ function as defined by the following criteria:

  1. ANC ≥ 1.5 × 10^9/L; excluding measurements obtained within 7 days after daily administration of filgrastim/sargramostim or within 3 weeks after administration of pegfilgrastim.
  2. Platelet count ≥ 100 × 10^9/L; excluding measurements obtained within 3 days after transfusion of platelets or within 3 weeks after administration of platelet growth factors.
  3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 × upper limit of normal (ULN). If liver function abnormalities are due to underlying liver metastases, AST and ALT ≤ 5 x ULN.
  4. Total serum bilirubin ≤ 1.5 × ULN or ≤ 3 × ULN in the case of Gilbert's disease.
  5. Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 60 mL/min.

Exclusion Criteria:

* Histology of abdominal adenocarcinoma of unknown origin or diagnosis of a borderline ovarian tumor.
* Any of the following treatment interventions within the specified time frame prior to Cycle 1 Day 1:

  1. Major surgery within 28 days.
  2. Radiation therapy within 21 days.
  3. Autologous or allogeneic stem cell transplant within 3 months.

A serious illness or medical condition(s) including, but not limited to, the following:

1. Brain metastases that require immediate treatment or are clinically or radiographically unstable.
2. Myocardial impairment of any cause.
3. Significant gastrointestinal abnormalities.
4. Active or uncontrolled infection.
5. Any evidence of small bowel obstruction as determined by air/fluid levels on computed tomography (CT) scan, recent hospitalization for small bowel obstruction within 3 months prior to Cycle 1 Day 1, or recurrent paracentesis or thoracentesis within 6 weeks prior to Cycle 1 Day 1.

   * Subjects with active (uncontrolled, metastatic) second malignancies or requiring therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
To investigate the safety and tolerability of ZN-c3 in combination with PLD, carboplatin, paclitaxel, gemcitabine, or bevacizumab | Through completion, approximately 40 months
  Incidence and severity of adverse events (AEs), graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0
To identify the maximum tolerated dose (MTD)/recommended Phase 2 dose (RP2D) of ZN-c3 in combination with PLD, carboplatin, paclitaxel, or gemcitabine | Through Cycle 1 (cycle is 28 days for PLD or paclitaxel, and 21 days for carboplatin, gemcitabine, or bevacizumab)
  Incidence and severity of dose-limiting toxicities (DLTs) in DLT-evaluable subjects during Cycle 1

CONTACTS AND LOCATIONS:
Locations (24):
- United States (8):
  - Site 0264, Aurora, Colorado
  - Site 0104, Boston, Massachusetts
  - Site 0111, St Louis, Missouri
  - Site 0173, New York, New York
  - Site 0259, Durham, North Carolina
  - Site 0191, Providence, Rhode Island
  - Site 0196, Nashville, Tennessee
  - Site 0103, Houston, Texas
- Australia (6):
  - Site 2707, South Brisbane, Queensland
  - Site 2708, Sunshine Coast, Queensland
  - Site 2709, Adelaide, South Australia
  - Site 2716, Melbourne, Victoria
  - Site 2706, Melbourne, Victoria
  - Site 2705, Nedlands, Western Australia
- Bosnia and Herzegovina (3):
  - Site 1001, Banja Luka
  - Site 1002, Sarajevo
  - Site 1003, Tuzla
- Bulgaria (2):
  - Site 1202, Panagyurishte
  - Site 1201, Sofia
- Site 1401, Tbilisi, Georgia
- Site 1902, Belgrade, Serbia
- South Korea (3):
  - Site 2901, Busan
  - Site 2903, Seoul
  - Site 2904, Seoul

IPD SHARING:
Plan to Share IPD: No